CLINICAL TRIAL: NCT02841670
Title: Evaluation of Efficacy and Long-term Safety for the InFo - Instant Focus © Lens / PMCF
Acronym: INFOLO
Status: Completed | Type: Observational
Sponsor: SAV-IOL SA (Industry)
Collaborators: CEISO (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-00909
Record Dates: First submitted 2016-07-12; First posted 2016-07-22 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: InFo - Instant Focus (c) lens implantation

SUMMARY:
This is a monocentric, longitudinal, prospective, observational post-market follow-up study.

30 patients with a cataract will receive an InFo - Instant Focus © lens implant. After the cataract procedure, data collection will take place during visits planned by the physician as part of normal follow-up.

Patients with cataract will be recruited from the clinic by the investigator based on the inclusion and exclusion criteria.

The patient will be followed up after one day, one week, one month, six months, one year and three years post-op. An interim analysis will be performed with one-year clinical results.

The main objective of the study is to evaluate is to evaluate efficacy and long-term safety for the InFo - Instant Focus © lens.

ELIGIBILITY:
Inclusion criteria:

* Suffering from cataract
* Physician has made the decision to implant on InFo - Instant Focus © lens
* Age ≥ 18 years, of either sex
* Having given written informed consent, prior to any procedure

Non inclusion criteria:

* Presenting with an astigmatism of >1.00D
* Presenting contraindications for the implantation of an intraocular lens
* Presenting an ophthalmic disorder liable to interfere with study endpoints
* History of previous intraocular surgery in the study eye in the previous 6 months
* Refusing or unable to comply with the follow-up schedule
* Participation in other interventional therapeutic trial at time of inclusion
* Pregnant, breastfeeding, or unable to understand the character and individual consequences of the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cataract will be recruited from the clinic by the investigator based on the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Near best corrected visual acuity | Year 1
Intermediate (80cm) best corrected visual acuity | Year 1
Far best corrected visual acuity | Year 1
Near uncorrected visual acuity | Year 1
Intermediate (80cm) uncorrected visual acuity | Year 1
Far uncorrected visual acuity | Year 1

SECONDARY OUTCOMES:
Contrast sensitivity | Year 1
Tilting sensitivity | Year 1
Decentration sensitivity | Year 1
Patient satisfaction | Year 1
  Questionnaire
Adverse events | Year 1
  Including Posterior Capsule Opacification rates

CONTACTS AND LOCATIONS:
Overall Officials: André Mermoud, Prof, Principal Investigator — Clinique Montchoisi Lausanne

IPD SHARING:
Plan to Share IPD: No